CLINICAL TRIAL: NCT03237910
Title: AMplitude Spectrum Area to Guide Defibrillation During Cardiopulmonary Resuscitation in Out-of-hospital Cardiac Arrest Patients
Brief Title: Real Time Amplitude Spectrum Area to Guide Defibrillation
Acronym: AMSA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: low rate recruitment
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Collaborators: European Commission (Other); Zoll Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRFMN-7167-7429
Record Dates: First submitted 2017-07-21; First posted 2017-08-03 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2021-09

CONDITIONS: Out-Of-Hospital Cardiac Arrest; Ventricular Fibrillation
Keywords: amplitude spectrum area; defibrillation; waveform analysis; cardiopulmonary resuscitation; cardiac arrest
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest; Ventricular Fibrillation; Heart Arrest | interventions — Electric Countershock; Cardiopulmonary Resuscitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- AMSA-CPR (Experimental): The professional rescuer decides to deliver the defibrillation attempt based on the AMSA value displayed in the defibrillator
  Interventions: Diagnostic Test: AMSA; Procedure: Defibrillation; Procedure: CPR
- Standard-CPR (Active Comparator): The defibrillation is delivered based on the 2015 European Resuscitation Council CPR guidelines
  Interventions: Procedure: Defibrillation; Procedure: CPR

INTERVENTIONS:
Diagnostic Test: AMSA — A non-invasive and real time VF (Amplitude Spectrum Area) AMSA analysis is performed during chest compression pauses for delivery of 2 ventilations, from the ECG acquired from the conventional defibrillatory pads
  Other Names: VF waveform analysis
  Arms: AMSA-CPR
Procedure: Defibrillation — delivery of the defibrillation is attempted to terminate VF either based on AMSA value (in the AMSA-CPR arm) or every 2-min CPR cycle as recommended by current guidelines (in the Standard-CPR arm)
  Other Names: electric countershock
Procedure: CPR — chest compressions and ventilations at a rate of 30:2
  Other Names: resuscitation maneuvres

SUMMARY:
AMSA trial is a multicenter, randomized, controlled study in out-of-hospital cardiac arrest patients.

The purpose of the study is to test the hypothesis that a real time AMSA analysis during CPR may predict the success of defibrillation and optimize the timing of defibrillation delivery.

The primary end-point is the efficacy of the AMSA-CPR: termination of VF/VT with achievement of ROSC for an AMSA ≥ 15.5 mV-Hz

All patients meeting inclusion/exclusion criteria and receiving cardiopulmonary resuscitation are randomized into two groups: AMSA-guided CPR or standard CPR.

In the AMSA-CPR group, AMSA value suggests when the rescuer should deliver the defibrillation attempt; In the Standard-CPR group, the defibrillation is delivered based on the 2015 European Resuscitation Council (ERC) CPR guidelines.

DETAILED DESCRIPTION:
In the AMSA-CPR intervention, upon arrival of the advanced life support (ALS) rescue team at the cardiac arrest scene and application of the defibrillatory pads to the patient's chest and power on of the defibrillator with the real time AMSA analysis:

* If AMSA is ≥ 15.5 mV-Hz, an immediate defibrillation is attempted, followed by CPR
* If AMSA is < 15.5 mV-Hz, defibrillation is not attempted and CPR is delivered
* During the 2-min cycle of CPR, AMSA is measured during pauses for ventilations (every 30 CC, approximately every 20/25 sec). If an AMSA value ≥ 15.5 mV-Hz is achieved prior to cycle completion, an immediate defibrillation is delivered (thus the defibrillation attempt is anticipated)

After completion of the first 2-min CPR cycle:

* If AMSA is ≤ 6.5 mV-Hz, the defibrillation is not attempted but CPR is continued
* If AMSA is > 6.5 mV-Hz, an immediate defibrillation attempt is delivered, followed by CPR
* During the 2-min cycle of CPR, AMSA is measured during pauses for ventilations (every 30 CC, approximately every 20/25 sec). If an AMSA value ≥ 15.5 mV-Hz is achieved prior to cycle completion, an immediate defibrillation is delivered

After completion of the second 2-min CPR cycle and till the end of the resuscitative intervention:

• CPR is continued based on standard 2015 ERC guidelines (a defibrillation attempt every 2-min CPR cycles), except for the possibility to anticipate the defibrillation attempt if AMSA becomes ≥ 15.5 mV-Hz during the CPR cycle.

In the standard CPR intervention, upon arrival of the ALS team at the cardiac arrest scene, and application of the defibrillatory pads to the patient's chest and power on of the defibrillator:

• a defibrillation is immediately attempted and CPR is then started and continued for 2- min. Analysis of rhythm and subsequent defibrillation attempts are performed every 2-min CPR cycles.

In both study groups, the quality of CC and ventilation is monitored in real time thought the feedback integrated into the defibrillator.

ELIGIBILITY:
Inclusion Criteria:

All adult patients (age ≥ 18) suffering of out-of-hospital non traumatic cardiac arrest of presumably cardiac etiology with a presenting shockable rhythm requiring electrical defibrillation: Ventricular Fibrillation and pulseless Ventricular Tachycardia.

Exclusion Criteria:

* age < 18 years old
* pregnancy
* cardiac arrest with a non-shockable rhythm (pulseless electrical activity and asystole)
* a defibrillation delivered by an AED prior to ALS arrival
* cardiac arrest of traumatic origin
* non-cardiac cause of cardiac arrest
* presumable irreversible death or known terminal illness at the beginning of ALS
* clinical death
* participation in another clinical or device trial within the previous 30 days
* refused informed consent to the use of data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2019-04-28 (Actual); Primary Completion 2021-07-26 (Actual); Study Completion 2021-07-26 (Actual)

PRIMARY OUTCOMES:
Return of spontaneous circulation (ROSC) | At day 0: from date of initiation of the cardiopulmonary resuscitation (CPR) maneuvres up to ROSC or up to 1 hour of CPR (which comes first)
  Termination of ventricular fibrillation with achievement of ROSC for an AMSA value ≥ 15.5 mV-Hz

SECONDARY OUTCOMES:
Defibrillation attempts | At day 0: from date of initiation of the cardiopulmonary resuscitation (CPR) maneuvres up to ROSC or up to 1 hour of CPR (which comes first)
  Number of defibrillations to achieve ROSC
CPR duration | At day 0: from date of initiation of the cardiopulmonary resuscitation (CPR) maneuvres up to ROSC or up to 1 hour of CPR (which comes first)
  duration of CPR in minutes prior to achieve ROSC
Cardiac troponins | at 6 and 24 hours after ICU admission
  assessment of circulating levels of high sensitive cardiac troponin T in plasma as marker of cardiac injury
Short term survival | at hospital admission and 24 hours after ROSC
  number of patients alive after initial resuscitation
Long term survival | at 1 and 6 months after ROSC
  number of patients alive after initial resuscitation

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Ristagno, MD, PhD, Study Chair — Istituto Di Ricerche Farmacologiche Mario Negri; Roberto Latini, MD, Study Chair — Istituto Di Ricerche Farmacologiche Mario Negri
Locations (2):
- Italy (2):
  - UOC Rianimazione-Emergenza Territoriale 118, Dipartimento di Emergenza, Ospedale Maggiore - AUSL di Bologna, Bologna
  - SOREU Metropolitana - AREU ASST, Grande Ospedale Metropolitano Niguarda, Milan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ruggeri L, Fumagalli F, Bernasconi F, Semeraro F, Meessen JMTA, Blanda A, Migliari M, Magliocca A, Gordini G, Fumagalli R, Sechi G, Pesenti A, Skrifvars MB, Li Y, Latini R, Wik L, Ristagno G. Amplitude Spectrum Area of ventricular fibrillation to guide defibrillation: a small open-label, pseudo-randomized controlled multicenter trial. EBioMedicine. 2023 Apr;90:104544. doi: 10.1016/j.ebiom.2023.104544. Epub 2023 Mar 26. PMID 36977371
- See also: EU Framework Horizon 2020 Programme under grant agreement no. 733381: European Sudden Cardiac Arrest network: towards Prevention, Education and New Treatment (ESCAPE-NET) — http://cordis.europa.eu/project/rcn/207233_en.html
- See also: ESCAPE NET in ERC website — https://www.erc.edu/projects/escape-net